CLINICAL TRIAL: NCT06414889
Title: Protocol Title: Safety and Feasibility of Autologous CD34+ Hematopoietic Stem Cells Mobilization and Apheresis in Participants With RUNX1 Familial Platelet Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: RUNX1 Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-0799; NCI-2024-04300 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: RUNX1 Familial Platelet Disorder
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Biosimilar Pharmaceuticals; pegfilgrastim; Blood Component Removal; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous CD34+ Hematopoietic Stem Cells Mobilization and Apheresis (Experimental): On Days 1-5, participants will receive a Granulocyte colony-stimulating factor (G-CSF), such as filgrastim, as an injection or by vein over about 5 minutes.
  If the study doctor thinks it is needed, participants will also receive plerixafor as an injection under the skin on Day 5 (and 6, if you have 2 days of apheresis).
  Interventions: Drug: G-CSF (filgrastim or biosimilar); Procedure: Apheresis; Drug: Plerixafor

INTERVENTIONS:
Drug: G-CSF (filgrastim or biosimilar) — Given by IV or SC
  Other Names: FILGRASTIM SD/01
Procedure: Apheresis — Given by procedure
Drug: Plerixafor — Given by IV

SUMMARY:
To evaluate the safety and feasibility of collecting hematopoietic stem cells (HSC) in participants with RUNX1-FPD.

DETAILED DESCRIPTION:
Primary Objective:

- To evaluate the safety of harvesting HSCs in participants with RUNX1 FPD

Secondary Objective

- To evaluate the feasibility and other relevant information of collecting HSCs from participants with RUNX1 FPD

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria are eligible to be included in the study:

1. Are aged ≥ 18 to 75 years

   a. Once a favorable review of safety has been completed by the SMC in 3 participants aged ≥ 18 years, the study will be opened to participants aged ≥ 12 years.
2. Are willing and able to provide informed consent, as appropriate (either directly or through a legally authorized representative [LAR]), as described in Appendix 1, Section 13.1
3. Have a confirmed diagnosis of RUNX1 FPD, verified by a Clinical Laboratory Improvement Amendments (CLIA)-certified genetic sequencing report.
4. Clearance by apheresis team to proceed
5. Have systolic blood pressure ≤ 170 mm Hg and diastolic blood pressure ≤ 95 mmHg
6. Are eligible for HSCT per institution requirements
7. Have a Lansky (age < 16 years)/Karnofsky performance status of ≥ 70 (see Appendix 2, Section 13.2).
8. Are willing and able to comply with protocol-defined contraceptive requirements (see Appendix 3 Section 13.3)
9. Have a platelet count ≥ 50,000/μL for initiation of apheresis, assessed within 24 hours prior to the procedure, or, if < 50,000/μL are administered platelets on the day of the collection

   a. If the apheresis team decides that a central venous catheter (CVC) is to be placed, platelet count should be ≥ 50,000 prior to catheter placement.
10. Have hemoglobin ≥ 7.5 g/dL as assessed within 24 hours prior to the procedure

Exclusion Criteria:

Participants who meet any of the following criteria are excluded from the study:

1. Participants with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with obtaining informed consent or compliance with study procedures.
2. Have uncontrolled bleeding
3. Are using supplemental oxygen
4. Have known severe splenomegaly (≥ 20 cm)
5. Have a diagnosis of MDS or hematologic malignancies, as defined by WHO hematolymphoid tumor classification fifth edition (Khourey et al 2022) hematolymphoid tumor classification fifth edition (Khourey et al 2022)
6. Have recent prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ Note: Cancer treated with curative intent < 5 years previously may be allowed following approval from the study investigator. Cancer treated with curative intent > 5 years previously is allowed.
7. Have any prior or current myeloproliferative or a significant coagulation or immunodeficiency disorder
8. Have advanced liver disease, defined as any of the following:

   1. Persistent aspartate transaminase, alanine transaminase, or direct bilirubin value > 5× the upper limit of normal (ULN) at screening
   2. Screening prothrombin time (PT) or partial thromboplastin time (PTT) > 1.5× ULN
9. Have had prior HSCT or gene therapy
10. Have history of concomitant sickle cell disease
11. Have been treated with an investigational drug within 30 days of screening or 5 half-lives (whichever is longer)
12. Have a positive test result for HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV) at screening

    1. Participants with positive hepatitis B core antibody (HbcAb) and/or hepatitis B-e antibody (HbeAb) are eligible provided viral load is negative by quantitative polymerase chain reaction (qPCR).
    2. Participants who are positive for anti-hepatitis C antibody are eligible as long as they have a negative HCV viral load by qPCR.
13. Have a positive infectious disease panel at screening for human T-lymphotropic virus 1 or 2 (HTLV-1 and HTLV-2), or syphilis (rapid plasma 24 reagin [RPR])
14. Have clinically significant and active bacterial, viral, fungal, or parasitic infection at screening
15. Have a white blood cell (WBC) count < 2 × 109/L
16. Have a left ventricular ejection fraction < 45%
17. Have a screening estimated glomerular filtration rate < 60 mL/min/1.73 m2
18. Have a diagnosis of a significant psychiatric disorder that could seriously impede the ability to participate in the study
19. For women of childbearing potential: are pregnant or breastfeeding or lack adequate contraception
20. Are unable to comply with the study procedures, as assessed by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Chitra Hosing, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org